CLINICAL TRIAL: NCT06757595
Title: Retrospective Analysis of the Clinical Characteristics of Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20241223
Record Dates: First submitted 2024-12-25; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Retinal Vein Occlusion
Keywords: Retinal Vein Occlusion; clinical feature; therapy
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- rvo patients
- Initial onset and meeting the diagnostic criteria for RVO (including BRVO and CRVO)

SUMMARY:
To explore the clinical characteristics of patients with RVO, and to analyze the relationship between RVO and various underlying diseases, ocular conditions, lifestyle, imaging findings and treatment response. To systematically analyze the clinical data of patients with different types of RVO, further reveal the potential mechanism of its occurrence and development, and evaluate the efficacy and safety of different treatment methods, in order to provide more scientific basis for clinical treatment.

DETAILED DESCRIPTION:
To explore the clinical characteristics of patients with RVO, and to analyze the relationship between RVO and various underlying diseases, ocular conditions, lifestyle, imaging findings and treatment response. To systematically analyze the clinical data of patients with different types of RVO, further reveal the potential mechanism of its occurrence and development, and evaluate the efficacy and safety of different treatment methods, in order to provide more scientific basis for clinical treatment.

Patients discharged from our hospital from January 2018 to December 2024 with the diagnosis of retinal vein occlusion were retrospectively investigated. The medical history of each patient was reviewed, and the basic information, past medical history, eye examinations and their results, treatment plans, and prognosis information of the patients were recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria for RVO (including BRVO and CRVO)

Exclusion Criteria:

* patients with other ocular diseases other than RVO, such as iridocyclitis, age-related macular degeneration, central serous chorioretinopathy and optic neuropathy;
* patients with systemic inflammatory diseases and other systemic diseases other than diabetes, hypertension, coronary heart disease and cerebral infarction that may affect blood indexes;
* patients with incomplete clinical data and information.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RVO diagnosed by ophthalmic examination in the Second Clinical Hospital of Wuhan University from January 2018 to December 2024 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Various underlying diseases, eye conditions, lifestyle, blood test results, imaging manifestations and treatment response | From January 2024 to January 2025
  Age, gender, blood routine (platelet count, neutrophil count, monocyte count, and lymphocyte count), four coagulation tests (prothrombin time determination, activated partial thromboplastin time determination), blood lipid (total cholesterol, triglyceride, high density lipoprotein, low density lipoprotein data), hypertension, diabetes, coronary heart disease, and cerebral infarction were collected in detail Death history, laser, anti-VEGF injection, hormone and other treatment methods and times, and the visual acuity at the last follow-up. The general conditions of the patients were statistically analyzed, such as the proportion of previous history of hypertension and diabetes, and the mean value of blood lipids, blood clotting images and other blood test results of the patients were calculated, and the correlation between them and the prognosis of vision was analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China